CLINICAL TRIAL: NCT04705376
Title: Cryotherapy Following Rotator Cuff Repair Surgery
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Funding
Sponsor: University Hospitals Cleveland Medical Center (Other)
Collaborators: Innovative Medical Equipment, LLC (Unknown); Ohio Third Frontier (Other)
Responsible Party: Principal Investigator, Robert J. Gillespie, Chief, Shoulder and Elbow Surgery, UH Cleveland Medical Center Program Director, Orthopaedic Surgery, UH Cleveland Medical Center Associate Professor, CWRU School of Medicine, University Hospitals Cleveland Medical Center
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: STUDY20200700
Record Dates: First submitted 2021-01-08; First posted 2021-01-12 (Actual); Last update posted 2022-04-22 (Actual); Status verified 2022-04

CONDITIONS: Rotator Cuff Tears
Keywords: Arthroscopy; Opioid Use
MeSH Terms: conditions — Rotator Cuff Injuries

STUDY DESIGN:
Intervention Model Description: The investigators propose a randomized crossover trial involving the use cryotherapy machines as a means of pain control following arthroscopic rotator cuff repair surgery. Patients will be randomized into receiving one of two possible cryotherapy devices immediately after surgery: Breg Polarcare or Thermazone. Randomization will occur with the use of a randomization excel spreadsheet. On post-operative day 3, patients who were originally randomized to Breg will then use Thermazone and patients who were randomized to Thermazone will use Breg for post-operative days 3 and 4. Both groups will alternate between both cryotherapy devices every two days post-operatively for 8 days total. Both groups will maintain a pain journal during the 8 study days post-operatively to document VAS scores, number of narcotic pain medications taken, and any adverse reactions from the cryotherapy devices. At 2 and 6-weeks follow-up, both groups will complete a functional evaluation.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Breg Polarcare (Active Comparator): Patients within the Breg Polarcare treatment arm will use the Breg Polarcare device for the first two days post-operatively following their arthroscopic rotator cuff repair. They will switch to the Thermazone device for post-operative days 3 and 4. They will continue to alternate every two days for 8 days total post-operatively.
  Interventions: Device: Breg Polarcare; Device: Thermazone
- Thermazone (Experimental): Patients within the Thermazone treatment arm will use the Thermazone device for the first two days post-operatively following their arthroscopic rotator cuff repair. They will switch to the Breg Polarcare device for post-operative days 3 and 4. They will continue to alternate every two days for 8 days total post-operatively.
  Interventions: Device: Breg Polarcare; Device: Thermazone

INTERVENTIONS:
Device: Breg Polarcare — The Breg Polarcare device is a type of cryotherapy machine that circulates ice cold water into a patch that can be worn by the patient on their affected joint (e.g., shoulder, knee).
Device: Thermazone — ThermaZone is a compact device that uses thermoelectric technology to provide heating and cooling therapy without the use of ice.

SUMMARY:
The purpose of this prospective crossover study is to determine if noninferiority exists in the use of the Thermazone cryotherapy machine when compared to Breg Polarcare, the current standard-of-care cryotherapy machine, for control of pain and reduction in postoperative narcotic medication consumption following arthroscopic rotator cuff repair surgery. Specifically, the investigators propose to test the hypothesis that in adults having arthroscopic rotator cuff repairs, the Thermazone device is non-inferior to Breg Polarcare on postoperative pain and opioid use over the initial 8 postoperative days.

DETAILED DESCRIPTION:
Cryotherapy has traditionally been used for the acute treatment of musculoskeletal injuries and following operative procedures. Cryotherapy currently represents the standard of care following common orthopaedic procedures to the knee and shoulder. In addition to relieving pain and swelling during the acute inflammatory period following surgery, cryotherapy has also been shown to reduce muscle spasms, promoting quicker functional recovery, accelerating post-operative rehabilitation and return to regular activities. Multiple investigations have demonstrated the benefit of cryotherapy following both shoulder and knee surgeries when compared to ice alone or no cryotherapy, however conflicting data prevents consensual agreement regarding the success of cryotherapy when compared to other post-operative pain control modalities.

The use of cryotherapy has been extensively studied in the shoulder following operative procedures. Kraeutler et al. compared compressive cryotherapy versus ice alone, reporting no reduction in pain between the two modalities following arthroscopic rotator cuff repair or subacromial decompression. Singh et al. reported in their randomized controlled trial that patients undergoing arthroscopic procedures to the shoulder reported lower pain intensity on Days 1, 14 and 21 with the use of cryotherapy compared to patients in the non-cryotherapy group. Meanwhile, Speer et al. found in their prospective study that use of cryotherapy in the post-operative period was associated with reduced pain and swelling, decreased opioid use and better sleep quality following arthroscopic rotator cuff repair.

Similar results have been reported in patients treated with cryotherapy following anterior cruciate ligament reconstruction. Seacrist et al. performed a systematic review, identifying 10 randomized controlled trials investigating the effects of cryotherapy/compression on pain management following anterior cruciate ligament reconstruction. Cryotherapy was found to improve analgesia compared to patients treated without cryotherapy in 4 trials, while in 4 trials ice water and water at room temperature provided equivalent analgesic effects. Raynor et al. found in their meta-analysis that cryotherapy following anterior cruciate ligament reconstruction significantly improved post-operative pain control, while no improvements in postoperative range of motion or drainage were appreciated. Meanwhile, a combined cryotherapy-compression device was found to result in a significantly higher percentage of patients discontinuing narcotics 6 weeks post-operatively with a significantly greater decrease in VAS scores from pre-operative levels at 2 and 6 weeks post-operatively when compared to ice packs alone.

Adverse reactions to cryotherapy including frostbite, cutaneous necrosis and neuropathy are rare, but have been reported, necessitating the need for appropriate use guidelines, recognition and prevention.

As such, despite multiple studies examining the post-operative impact of cryotherapy following shoulder and knee procedures, no definitive conclusions on the effectiveness of cryotherapy on outcomes related to the use of post-operative analgesic medication, pain control, functional outcomes and range of motion have been determined. The conflicting reports regarding the benefit of cryotherapy may be related to the failure to achieve required decreases in intra-articular temperatures. Additional investigations are needed to better understand the impact of cryotherapy following arthroscopic rotator cuff, shoulder labral repair, anterior cruciate ligament reconstruction and meniscal repair/resection procedures.

Breg polarcare is a commonly used cryotherapy device that has a variety of clinical applications. The polarcare device requires ice and water, which is then circulated through a pad which the patient applies directly to the affected area. The Thermazone device does not require the use of ice and allows for osscilation between hot and cold temperatures. Currently, both cryotherapy devices are approved for use following surgery. However, no study to date has compared the Breg polarcare and thermazone devices in the context of arthroscopic rotator cuff surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing primary arthroscopic rotator cuff repair.

Exclusion Criteria:

* Patients with any of the following pre-existing medical conditions: Fibromyalgia; Complex regional pain syndrome; Any pain disorder that requires the patient to take narcotic pain medication in the pre-operative time period
* Patients undergoing revision arthroscopic rotator cuff surgery
* Illiterate, non-English speaking, and pregnant individuals

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2021-09-01 (Estimated); Study Completion 2021-11-01 (Estimated)

PRIMARY OUTCOMES:
Pain Visual Analog Scale | 2 weeks post-operatively
  Scale from 0 to 10; 0 represents no pain and 10 represents the most amount of pain.
Pain Visual Analog Scale | 6 weeks post-operatively
  Scale from 0 to 10; 0 represents no pain and 10 represents the most amount of pain.
American Shoulder and Elbow Surgeons (ASES) Score | 2 weeks post-operatively
  Scale from 0 to 100 with higher scores representing better outcomes. The total score is weighted 50% for pain and 50% for function.
American Shoulder and Elbow Surgeons (ASES) Score | 6 weeks post-operatively
  Scale from 0 to 100 with higher scores representing better outcomes. The total score is weighted 50% for pain and 50% for function.
Simple Shoulder Test (SST) | 2 weeks post-operatively
  Scale ranges from 0% to 100% with higher scores representing better outcomes. Consists of a series of 12 "yes" or "no" questions the patient answers about the function of the involved shoulder. The answers to these questions provides a standardized way of recording the function of a shoulder before and after treatment.
Simple Shoulder Test (SST) | 6 weeks post-operatively
  Scale ranges from 0% to 100% with higher scores representing better outcomes. Consists of a series of 12 "yes" or "no" questions the patient answers about the function of the involved shoulder. The answers to these questions provides a standardized way of recording the function of a shoulder before and after treatment.

SECONDARY OUTCOMES:
Adverse reactions from cryotherapy devices | 2 weeks post-operatively
  The investigators will assess the rate of adverse reactions from the two cryotherapy devices and develop and adverse reaction profile.
Adverse reactions from cryotherapy devices | 6 weeks post-operatively
  The investigators will assess the rate of adverse reactions from the two cryotherapy devices and develop and adverse reaction profile.

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospitals Cleveland Medical Center, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Khoshnevis S, Craik NK, Diller KR. Cold-induced vasoconstriction may persist long after cooling ends: an evaluation of multiple cryotherapy units. Knee Surg Sports Traumatol Arthrosc. 2015 Sep;23(9):2475-83. doi: 10.1007/s00167-014-2911-y. Epub 2014 Feb 23. PMID 24562697
- [Background] Kraeutler MJ, Reynolds KA, Long C, McCarty EC. Compressive cryotherapy versus ice-a prospective, randomized study on postoperative pain in patients undergoing arthroscopic rotator cuff repair or subacromial decompression. J Shoulder Elbow Surg. 2015 Jun;24(6):854-9. doi: 10.1016/j.jse.2015.02.004. Epub 2015 Mar 29. PMID 25825138
- [Background] Raynor MC, Pietrobon R, Guller U, Higgins LD. Cryotherapy after ACL reconstruction: a meta-analysis. J Knee Surg. 2005 Apr;18(2):123-9. doi: 10.1055/s-0030-1248169. PMID 15915833
- [Background] Secrist ES, Freedman KB, Ciccotti MG, Mazur DW, Hammoud S. Pain Management After Outpatient Anterior Cruciate Ligament Reconstruction: A Systematic Review of Randomized Controlled Trials. Am J Sports Med. 2016 Sep;44(9):2435-47. doi: 10.1177/0363546515617737. Epub 2015 Dec 18. PMID 26684664
- [Background] Song M, Sun X, Tian X, Zhang X, Shi T, Sun R, Dai W. Compressive cryotherapy versus cryotherapy alone in patients undergoing knee surgery: a meta-analysis. Springerplus. 2016 Jul 13;5(1):1074. doi: 10.1186/s40064-016-2690-7. eCollection 2016. PMID 27462522
- [Background] Speer KP, Warren RF, Horowitz L. The efficacy of cryotherapy in the postoperative shoulder. J Shoulder Elbow Surg. 1996 Jan-Feb;5(1):62-8. doi: 10.1016/s1058-2746(96)80032-2. PMID 8919444
- [Background] Uquillas CA, Capogna BM, Rossy WH, Mahure SA, Rokito AS. Postoperative pain control after arthroscopic rotator cuff repair. J Shoulder Elbow Surg. 2016 Jul;25(7):1204-13. doi: 10.1016/j.jse.2016.01.026. Epub 2016 Apr 11. PMID 27079219
- [Background] Waterman B, Walker JJ, Swaims C, Shortt M, Todd MS, Machen SM, Owens BD. The efficacy of combined cryotherapy and compression compared with cryotherapy alone following anterior cruciate ligament reconstruction. J Knee Surg. 2012 May;25(2):155-60. doi: 10.1055/s-0031-1299650. PMID 22928433
- [Background] Tashjian RZ, Shin J, Broschinsky K, Yeh CC, Martin B, Chalmers PN, Greis PE, Burks RT, Zhang Y. Minimal clinically important differences in the American Shoulder and Elbow Surgeons, Simple Shoulder Test, and visual analog scale pain scores after arthroscopic rotator cuff repair. J Shoulder Elbow Surg. 2020 Jul;29(7):1406-1411. doi: 10.1016/j.jse.2019.11.018. Epub 2020 Feb 17. PMID 32081634
- [Background] Singh H, Osbahr DC, Holovacs TF, Cawley PW, Speer KP. The efficacy of continuous cryotherapy on the postoperative shoulder: a prospective, randomized investigation. J Shoulder Elbow Surg. 2001 Nov-Dec;10(6):522-5. doi: 10.1067/mse.2001.118415. PMID 11743529